CLINICAL TRIAL: NCT05489250
Title: The Platform for Analyzing Targetable Tumor Mutations Network (Main-study)
Brief Title: The PLATON Network
Acronym: PLATON
Status: Terminated | Type: Observational
Why Stopped: Sponsor Decision
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Other Study IDs: The PLATON Network
Record Dates: First submitted 2022-05-31; First posted 2022-08-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hepatocellular Cancer; Cholangiocarcinoma; Gallbladder Cancer; Pancreatic Cancer; Oesophageal Cancer; Stomach Cancer
Keywords: Gastric cancer; Individualized cancer therapy; Targetable mutations; NGS; Hepatocellular Cancer; Cholangiocarcinoma; Gallbladder Cancer; Pancreatic Cancer; Oesophageal Cancer; Stomach Cancer; Platform-Design; Biobanking
MeSH Terms: conditions — Liver Neoplasms; Cholangiocarcinoma; Gallbladder Neoplasms; Pancreatic Neoplasms; Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum and plasma, formalin-fixed paraffin-embedded tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HCC (Hepatocellular cancer): Hepatocellular cancer patients with NGS based molecular tumor profiling
- CCA/GBCA (Intra-, extrahepatic cholangiocellular carcinoma or gallbladder cancer): Intra-, extrahepatic cholangiocellular carcinoma or gallbladder cancer patients with NGS based molecular tumor profiling
- PanCa (Pancreatic cancer): Pancreatic cancer patients with NGS based molecular tumor profiling
- EC/GC (Oesophagogastric cancer): Oesophagogastric cancer patients with NGS based molecular tumor profiling

SUMMARY:
The PLATON Network study is designed to elevate personalized therapy based on genomic tumor profiles in gastrointestinal cancer patients. Hereby, PLATON's study-design focuses on the patient's tumor molecular profiling. Within the network a web application will be developed to link clinical investigators and information on study sites, cancer patients and genetic alteration data, as well as available clinical trials at PLATON's study sites.

DETAILED DESCRIPTION:
The PLATON Network is established as permanent open, multicenter, prospective, cohort study of patients with gastrointestinal cancer. The study design includes a study-specific biobank and a shared platform infrastructure for associated sub-studies and analysis projects.

Within PLATON results of genetic tests of different research projects like the PLATON pilot-study (NCT04484636) as well as Next-generation deep sequencing (NGS) according to local protocols will be documented - compiling genomic tumor-profiles including tumor mutational burden (TMB) and microsatellite instability (MSI).

The PLATON Network infrastructure is designed to increase the likelihood of treating the patients with an individualized therapy in available clinical studies. Therefore, molecular profiling must go hand in hand with inter-linking physicians and increasing inter-centre transparency. The feasibility of this approach will be tested in the PLATON Network, keeping in mind the vision of cancer patients receiving the best available, scientifically founded, biomarker-based care, tailored to his or her individual needs.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of hepatocellular carcinoma or intra- cholangiocarcinoma, extrahepatic cholangiocarcinoma or gallbladder carcinoma or pancreatic ductal adenocarcinoma or esophagogastric adenocarcinoma in the advanced setting (adjuvant or neoadjuvant therapy is allowed if completed 6 months prior to enrolment) and no local curative therapy available
* Standard first line therapy is planned, or patient is currently receiving first-line therapy
* Available tumor-genomic profile ( ≥50-gene panel assay; approved and assessed by central review), unless central tumor genomic profiling is done within a sub-study
* ECOG 0-2
* Life expectancy ≥ 6 months

Exclusion Criteria:

* Not able to understand all implications of study participation
* No written informed consent
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The PLATON Network and its associated pilot study (clinicaltrials.gov:. NCT04484636) enrolls national-wide participants of both sexes and ages over 18 years. All participants are patients diagnosed with hepatocellular cancer (HCC) or intra-/extrahepatic cholangiocellular carcinoma (CCA) or gallbladder carcinoma (GBCA) or pancreatic cancer (PanCa) or esophagogastric cancer (EC/GC). At the time of enrolment life expectancy is at least 6 months and no local curative therapy is available.
Sampling Method: Probability Sample
Enrollment: 565 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Frequency of targetable mutations in gastrointestinal cancer patients | annual interim-analysis (1 year)
  Relative frequency of targetable mutations computed as the number of patients who harbor at least one mutation divided by the number of total patients in the analyzed patient population
Tumor mutations and their impact on treatment decisions in gastrointestinal cancer patients | annual interim-analysis (1 year)
  Number of received therapies in or out accordance to genomic profiles

SECONDARY OUTCOMES:
Overall survival (OS) in genetically defined cohorts in gastrointestinal cancer patients | annual interim-analysis (1 year)
  Overall survival measurement over time grouped by diagnostic cohorts and adjusted by age and sex will be correlated to treatments, while genomic profiles had or had not impact on decision for treatment.
QoL via EQ-5D-5L questionnaire in genetically defined cohorts in gastrointestinal cancer patients | annual interim-analysis (1 year)
  QoL measurements are done over time in the palliative setting. Gastrointestinal cancer patient cohorts will be grouped by diagnostics and adjusted by age and sex, correlated to treatments, while genomic profiles had or had not impact on decision for treatment in gastrointestinal cancer patients.
  EQ-5D data is used in summary statistics at each observational timepoint and to estimate the difference between health states like "Mobility", "Looking After Myself", "Doing Usual Activities", "Having Pain or Discomfort", "Feeling Worried, Sad or Unhappy" in diagnostic groups of different treatments over time. The EQ VAS (visual analogue scale) on a scale from 0 (the worst imaginable health) to 100 (the best imaginable health) indicates patients´ overall health on the day of questionnaire completion and will be used as measure of central tendency and dispersion
QoL via EORTC QLQ-C30 questionnaire in genetically defined cohorts in gastrointestinal cancer patients | annual interim-analysis (1 year)
  QoL measurements are done over time in the palliative setting. Gastrointestinal cancer patient cohorts will be grouped by diagnostics and adjusted by age and sex, correlated to treatments, while genomic profiles had or had not impact on decision for treatment in gastrointestinal cancer patients.
  EORTC QLQ-C30 data is used in summary statistics at each observational timepoint to analyze five function subscales (physical, role, emotional, cognitive and social), nine symptom subscales/items (fatigue, nausea/vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhoea and financial difficulties) and a global health/ QoL subscale following the QLQ-C30 scoring manual.
QoL via EORTC QLQ-BIL21 questionnaire in genetically defined cohorts of CCA and GBCA patients | annual interim-analysis (1 year)
  QoL measurements are done over time in the palliative setting. The CCA and GBCA patients cohort will be adjusted by age and sex, correlated to treatments, while genomic profiles had or had not impact on decision for treatment.
  QoL in CCA and GBCA patients will be measured using the European Organisation for Research and Treatment of Cancer (EORTC) Questionnaire QLQ-BIL21 and analyzed according validated manual, forming nine symptom subscales/items for "Eating", "Jaundice", "Tiredness", "Pain" and "Anxiety".
QoL via EORTC QLQ-HCC18 questionnaire in genetically defined cohorts of HCC patients | annual interim-analysis (1 year)
  QoL measurements are done over time in the palliative setting. The HCC patient cohort will be adjusted by age and sex, correlated to treatments, while genomic profiles had or had not impact on decision for treatment.
  QoL in HCC patients will be measured using the European Organisation for Research and Treatment of Cancer (EORTC) Questionnaire QLQ-HCC18 and analyzed according validated manual, forming symptom scales for "Fatigue", "Body Image", "Jaundice", "Nutrition", "Pain" and "Fever" as well as single items like "Abdominal swelling" and "Sex life" in summary statistics at each observational timepoint.
QoL via EORTC QLQ-PAN26 questionnaire in genetically defined cohorts of PDCA patients | annual interim-analysis (1 year)
  QoL measurements are done over time in the palliative setting. The PDCA patient cohort will be adjusted by age and sex, correlated to treatments, while genomic profiles had or had not impact on decision for treatment.
  QoL in PDCA patients will be measured using the European Organisation for Research and Treatment of Cancer (EORTC) Questionnaire QLQ-PAN26 and analyzed according validated manual, forming eight scales to assess "Pancreatic pain", "Digestive symptoms", "Altered bowel habit", "Hepatic, body image", "Satisfaction with health care", and "Sex life" in summary statistics at each observational timepoint.
QoL via EORTC QLQ-STO22 questionnaire in genetically defined cohorts of EC/GC patients | annual interim-analysis (1 year)
  QoL measurements are done over time in the palliative setting. The EC/GC patient cohort will be adjusted by age and sex, correlated to treatments, while genomic profiles had or had not impact on decision for treatment.
  QoL in EC/GC patients will be measured using the European Organisation for Research and Treatment of Cancer (EORTC) Questionnaire QLQ-STO22 and analyzed according validated manual, forming five multi-item scales to assess "dysphagia", "pain", "reflux", "eating" and "anxiety" as well as four single items like "dry mouth", "taste", "body image" and "hair loss" in summary statistics at each observational timepoint.

OTHER OUTCOMES:
Feasibility of the PLATON WebApp - an interactive platform that connects the participating physicians on cases, cancer types, mutations, protein expressions and therapies, possible trials and discussion options for medical professionals | through study completion, an average of 2 years
  The feasibility will be analyzed with a usability questionnaire regarding user experience, design criteria etc. of the newly designed infrastructure and an additional count on possible matches of cancer patients with defined genetic tumor-profiles to possible targeted therapy strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof. Dr., Study Director — Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest; Arndt Vogel, Prof. Dr., Principal Investigator — Hannover Medical School (MHH)
Locations (31):
- Germany (31):
  - KHNW Frankfurt, Frankfurt am Main, Hesse
  - Friedrich-Ebert-Krankenhaus Neumünster, Neumünster, Schleswig-Holstein
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - Evangelisches Waldkrankenhaus Spandau, Berlin
  - MVZ Oskar-Helene-Heim Berlin, Berlin
  - Augusta-Kranken-Anstalt Bochum, Bochum
  - Bochum Uni, Bochum
  - Klinikum Chemnitz, Chemnitz
  - GEFOS - Gesellschaft für onkologische Studien Dortmund, Dortmund
  - Onkozentrum Dresden, Dresden
  - Ev. Kliniken Essen-Mitte, Klinik für Internistische Onkologie, Essen
  - MVZ Onkologische Kooperation Harz, Goslar
  - Universitätsklinikum Halle (Saale), Halle
  - Hamburg Onkologische Schwerpunktpraxis Eppendorf, Hamburg
  - St. Anna Hospital Herne, Herne
  - Ortenau Klinikum Lahr-Ettenheim, Lahr
  - ÜBAG - MVZ Dr. Vehling-Kaiser GmbH, Landshut
  - Langen, Gemeinschaftspraxis für Hämatologie und Onkologie, Langen
  - Studienzentrum UnterEms, Leer
  - Klinikum Lippe, Lemgo
  - Klinikum Ludwigsburg, Ludwigsburg
  - Klinik München-Bogenhausen, München
  - Münster, Gemeinschaftspraxis für Hämatologie und Onkologie, Münster
  - Medius Klinik Osterfildern-Ruit, Ostfildern
  - Krankenhaus Barmherzige Brüder, Regensburg
  - Klinikum Rheine, Mathias-Spital Rheine, Rheine
  - CaritasKlinikum Saarbrücken, Saarbrücken
  - Onkologie Bodensee, Singen
  - Marien Hospital Witten, Witten
  - Klinikum Wolfsburg, Wolfsburg
  - Onkologisches Zentrum Wolfsburg-Helmstedt MVZ GmbH, Wolfsburg

IPD SHARING:
Plan to Share IPD: Yes
Depending on participant informed consent individual-participant data (IPD) will be shared in research-cooperations according the terms of PLATON's Use and Access Regulation for scientific and/or educational use. Scientific/ educational projects have to be approved by PLATON'S Scientific Steering Committee.
Supporting Information: Study Protocol, ICF, CSR
Access Criteria: PLATON's Use und Access Regulation is available upon individual request for PLATON Network members and cooperation partners. For more information on contact please visit the PLATON Network website.
URL: https://platon-network.de/contact

REFERENCES:
- See also: The PLATON Network - website with study information (public) — https://platon-network.de/
- See also: The PLATON Network - PLATON WebApp (web-application for PLATON network members only) — http://platonwebapp.de
- See also: The PLATON Network - Data Capture (for PLATON study team members only) — https://asp.interactive-systems.de/cgi-bin/WebObjects/ST50-productive-DataCapture.woa/wa/choose?customer=TGO
- Available data/document: Informed Consent Form — https://platon-network.de/contact
- Available data/document: See Use & Access Regulation — https://platon-network.de/contact